CLINICAL TRIAL: NCT00464048
Title: A Controlled Study to Assess the Effectiveness of Aerobic Exercise as an Augmentation Therapy for Inpatients With Major Depressive Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: bhmi55-hmo-ctil
Record Dates: First submitted 2007-04-19; First posted 2007-04-20 (Estimated); Last update posted 2007-04-20 (Estimated); Status verified 2007-04

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: controlled physical exercise

SUMMARY:
We will evaluate the effect of a short-term aerobic exercise program as an adjuvant treatment in patients with depression undergoing standard clinical antidepressant medication therapy as compared to the effect of stretching exercise. In addition, the effect of exercise on plasma biological markers will be examined and observed changes correlated with clinical antidepressant effects. We hypothesize that the aerobic exercise group will achieve a significantly higher response rates of depressive symptoms, will also have a greater degree of change in the plasma markers, than the control stretching group.

DETAILED DESCRIPTION:
The patients will be randomly assigned to 3 weeks of augmentation therapy (in addition to the antidepressant medication, which will be continued) with either: 1) aerobic exercise or 2) stretching exercise (control group). Random assignment to each group will be stratified according to previous response to treatment as determined by a psychiatrist and review of the Antidepressant Treatment History Form (ATHF) and by gender.

Severity of depression will be rated at the first baseline visit and every week during the exercise program using the Hamilton Depression Scale (HAM-D 21 items), Clinical Global Impression Scale (CGI) (observer-rated) and Beck Depression Inventory (BDI) and Visual Analog Scale (self-rated).

Blood samples will be obtained four times during the study - before and after the first exercise session and before and after the last exercise session. The blood taken before the exercise sessions will be used to assay thyroxine, cortisol, insulin, opioid peptides and cytokines such as IL-6 and TNF-α in the plasma. The blood taken after the exercise sessions will be used to re-examine variables expected to be altered immediately after exercise such as cortisol, opioid peptides, catecholamines and cytokines.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Major Depressive Episode (MDE) in the context of MDD according to DSM-IV criteria, without psychotic features.
2. Hamilton Depression Scale (21 items, HAM-D) total>14 with item 1 (depressed mood) >2.
3. Physical capability to perform aerobic exercise or stretching exercise.
4. Competent and willing to give written informed consent

Exclusion Criteria:

1. Current, significant physical illness that will preclude exercise training.
2. Any physical impairment that can interfere with exercise training.
3. Current psychotic features.
4. Treatment with electroconvulsive therapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-05; Study Completion 2009-05 (Estimated)

PRIMARY OUTCOMES:
response of depressive symptoms- reduction in HAM-D score at the end of the follow-up period

SECONDARY OUTCOMES:
reduction in pretreatment BDI score
remission according to HAM-D score
remission according to BDI score
changes in plasmatic measurements before and after the first and last exercise
length of hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: tal Shahar, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel